CLINICAL TRIAL: NCT03502447
Title: Randomized, Controlled Trial to Evaluate the Safety and Effectiveness of the TearCare® System in the Treatment of the Signs and Symptoms of Dry Eye Disease
Brief Title: Randomized Study of the Safety and Effectiveness of the TearCare System for the Signs and Symptoms of Dry Eye Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor chose to change the study design.
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05474
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TearCare (Experimental): TearCare subjects will receive TearCare thermal treatment followed by manual clearing of the meibomian glands.
  Interventions: Device: TearCare
- Warm Compress & Lid Massage (Active Comparator): Subjects will perform warm compress and lid massage at home daily.
  Interventions: Device: Warm Compress and Lid Massage

INTERVENTIONS:
Device: TearCare — TearCare treatment includes an in-office 15 minute thermal treatment session where heat is delivered to the eyelids. This is immediately followed by manual clearing of the meibomian glands.
  Arms: TearCare
Device: Warm Compress and Lid Massage — Subjects randomized to the Warm Compress and Lid Massage Group will be instructed to apply a moist, warm compress to their eyelids daily for 5 minutes and then perform lid massage.
  Arms: Warm Compress & Lid Massage

SUMMARY:
In this study, the TearCare System will be compared with standard-of-care warm compress treatment and lid massage in patients with dry eye disease. The objective is to demonstrate that the TearCare System is safe and effective in relieving the signs and symptoms of dry eye disease and that it is superior to a commonly prescribed, standard treatment of warm compress and lid massage.

NOTE: All sites have been selected for this study.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, single-masked, multi-center treatment study will recruit 200 subjects with dry eye disease (OSDI Score of ≥23, TBUT of ≤7 seconds in both eyes, Meibomian gland obstruction in both eyes based on a total Meibomian Gland Secretion Score ≤12 in each eye and best corrected visual acuity of 20/100 or better in both eyes). Subject will be at least 22 years of age with reports of dry eye symptoms within the past 3 months, having to use artificial tears or lubricants regularly over the past month to relieve dry eye symptoms and willingness to comply with the study procedures and follow-up for 12 months.

All subjects will complete an informed consent form indicating their voluntary participation in the study.

Study Measurements will be made at baseline (Day 0 - randomization to TearCare or Warm Compress/Lid Massage) and at Day 1, Week 1, and Months 1, 3, 6, 7, 9, 12.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dry eye disease
* Signs and symptoms of dry eye disease
* Best corrected visual acuity 20/100 or better
* Willing and able to comply with study procedures
* Willing and able to provide consent

Exclusion Criteria:

* Active ocular infection or inflammation
* History of eyelid, conjunctiva or corneal surgery within the past year.
* Recent office-based dry eye treatment, punctal occlusion or punctal plug placement
* Contact lens wearer
* Significant ocular surface or eyelid abnormalities, recent ocular trauma
* Certain corneal surface abnormalities
* Use of medications for treatment of dry eye or medications that cause dry eye
* Systemic disease that results in dry eye

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Dickerson, PhD, Study Director — Sight Sciences, Inc.
Locations (6):
- United States (6):
  - Harvard Eye Associates, Laguna Hills, California
  - Eye Research Foundation, Newport Beach, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Ophthalmology Associates, St Louis, Missouri
  - Vance Thompson Vision, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TearCare | Warm Compress & Lid Massage
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TearCare | Warm Compress & Lid Massage | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10.1) | 55.9 (20.9) | 62.45 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Tear Break Up Time [Mean (Standard Deviation); unit: seconds] — The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit.
  seconds | 4.9 (0.8) | 4.7 (0.7) | 4.8 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Tear Break-Up Time From Baseline to Month 1
Description: The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit. The change in TBUT was The difference between the mean baseline value and the mean Month 1 value. The TBUT for each eye for a subject was averaged. The mean change in TBUT is the Month 1 value minus the baseline value for each subject which are then averaged. An increase in TBUT is an improvement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TearCare | Warm Compress & Lid Massage
Number analyzed (Participants) | 7 | 7
seconds | 1.4 (2.3) | 2.5 (2.8)

2. Secondary Outcome: Mean Change in OSDI Score From Baseline to Month 1
Description: The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire that assesses symptoms of ocular irritation associated with dry eye and the impact of these on vision-related activities. The OSDI score ranges from 0 (best possible) to 100 (worst possible). The change in OSDI questionnaire from baseline to Month 1 is the difference between the scores at the two timepoints. A negative value would indicate improvement and a positive value, a worsening. The reported value is the mean of the change for all subjects.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare | Warm Compress & Lid Massage
Number analyzed (Participants) | 7 | 7
units on a scale | -13.7 (12.5) | -10.0 (7.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All the study procedures meet non-significant risk criteria. Thus, no patients were at risk of either Serious Adverse Events or All-Cause Mortality.
  No adverse events noted from study start to early termination.
Arm/Group | TearCare | Warm Compress & Lid Massage
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03502447/Prot_SAP_002.pdf